CLINICAL TRIAL: NCT02278692
Title: Evaluation of Vitamin K Supplementation for Calcific Uremic Arteriolopathy
Acronym: VitK-CUA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Kidney Foundation, United States (Other); American Heart Association (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Sagar U. Nigwekar, MD, MMSc, Assistant Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014P001961
Record Dates: First submitted 2014-10-27; First posted 2014-10-30 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Calciphylaxis; Calcific Uremic Arteriolopathy
Keywords: Vitamin K; Calciphylaxis; Calcific uremic arteriolopathy; Dialysis; End-stage renal disease
MeSH Terms: conditions — Calciphylaxis; Kidney Failure, Chronic | interventions — Vitamin K

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin K (Active Comparator): Vitamin K1 (phytonadione) 10 mg orally three times a week after dialysis for 12 weeks
  Interventions: Dietary Supplement: Vitamin K
- Placebo (Placebo Comparator): Identical appearing placebo orally three times a week after dialysis for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin K — Oral vitamin K
  Arms: Vitamin K
Other: Placebo — Oral placebo tablet
  Arms: Placebo

SUMMARY:
Calcific uremic arteriolopathy a.k.a. calciphylaxis is a vascular calcification disorder seen in dialysis patients. Calcific uremic arteriolopathy has 60-80% one-year mortality and significant morbidity associated with non-healing and extremely painful skin lesions. At present, there is no effective treatment for calcific uremic arteriolopathy.

Vitamin K is an important vitamin for inhibiting vascular calcification. It is known to increase the circulating levels of carboxylated Matrix Gla Protein, a potent inhibitor of vascular calcification. However, the effects of vitamin K supplementation in patients with calcific uremic arteriolopathy are unknown.

The purpose of this study is to conduct a pilot randomized controlled trial to examine the effects of oral vitamin K supplementation on circulating levels of anti-calcification factor (carboxylated Matrix Gla Protein) and clinical outcomes in patients with calcific uremic arteriolopathy.

DETAILED DESCRIPTION:
Calcific uremic arteriolopathy (CUA), also known as calciphylaxis, is a vascular calcification disorder associated with 60-80% one-year mortality and significant morbidity. CUA predominantly affects end-stage renal disease (ESRD) patients and presents with painful skin lesions. Although rare (prevalence: 4% in dialysis patients), the incidence of CUA is on the rise as shown by us and others. Mural calcification of dermal arterioles is the hallmark histological finding of CUA. However, there are significant gaps in the understanding of the pathophysiology and risk factors for CUA and there are no effective therapies.

In animal models, vitamin K prevents vascular calcification by serving as a co-factor for Matrix Gla Protein (MGP) carboxylation, a process that converts decarboxylated-MGP (dc-MGP) to carboxylated-MGP (c-MGP). By inhibiting pro-calcification Bone Morphogenic Protein (BMP) ligands, c-MGP acts as a potent vascular calcification inhibitor. uc-MGP is inactive with no vascular calcification inhibitory properties. However, the effects of vitamin K administration on CUA remain unknown.

Aim: To conduct a pilot randomized controlled trial (RCT) of oral vitamin K in CUA.

The investigators will examine the following hypotheses:

Hypothesis 1: Vitamin K therapy, when compared to placebo, reduces uncarboxylated Matrix Gla Protein in chronic hemodialysis patients with CUA.

Hypothesis 2: Vitamin K therapy can be safely administered in chronic hemodialysis patients with CUA.

Hypothesis 3: Vitamin K therapy leads to improvement in CUA pain and average lesion size when compared to placebo in chronic hemodialysis patients.

Study population and procedures: Twenty patients will be enrolled in this pilot RCT over the 2-year study period.

Study Procedures: Patients meeting the eligibility criteria will be consented and randomized to receive either vitamin K (phylloquinone) 10 mg orally three times a week for a total of 12 weeks or identical appearing placebo. Follow-up will occur every 4 weeks during which information will be obtained regarding pain severity, number and size of CUA lesion (s), and adverse events. Blood samples will be taken at baseline and at 12-week follow-up.

Sample processing and assays: Blood samples (plasma and serum, total 30 mL) will be taken at baseline and at 12-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Calcific uremic arteriolopathy (a.k.a. calciphylaxis)

Exclusion Criteria:

* Warfarin discontinuation contra-indicated (e.g. mechanical heart valve)
* Prior allergic reaction to vitamin K
* Prior history of venous thromboembolism*
* Pregnancy and lactation

(*Patients with prior history of thrombosis who are treated with non-warfarin anticoagulant agents (e.g. apixaban, enoxaparin, etc) will be considered for inclusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-03; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in circulating MGP level at 12 weeks | Baseline and 12 weeks

SECONDARY OUTCOMES:
Change from baseline in largest lesion size at 12 weeks | Baseline and every month for 3 months
  Lesion size is measured in centimeters2
Change from baseline in combined area of all lesions at 12 weeks | Baseline and every month for 3 months
  Lesion size is measured in centimeters2
Change from baseline in pain at 12 weeks | Baseline and every month for 3 months
  Pain is measured using Wong-Baker Faces pain rating scale

OTHER OUTCOMES:
Adverse events | Baseline and every month for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Nigwekar, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Nigwekar SU, Brunelli SM, Meade D, Wang W, Hymes J, Lacson E Jr. Sodium thiosulfate therapy for calcific uremic arteriolopathy. Clin J Am Soc Nephrol. 2013 Jul;8(7):1162-70. doi: 10.2215/CJN.09880912. Epub 2013 Mar 21. PMID 23520041
- [Background] Nigwekar SU, Bhan I, Turchin A, Skentzos SC, Hajhosseiny R, Steele D, Nazarian RM, Wenger J, Parikh S, Karumanchi A, Thadhani R. Statin use and calcific uremic arteriolopathy: a matched case-control study. Am J Nephrol. 2013;37(4):325-32. doi: 10.1159/000348806. Epub 2013 Mar 21. PMID 23548843
- [Background] Nigwekar SU, Bloch DB, Nazarian RM, Vermeer C, Booth SL, Xu D, Thadhani RI, Malhotra R. Vitamin K-Dependent Carboxylation of Matrix Gla Protein Influences the Risk of Calciphylaxis. J Am Soc Nephrol. 2017 Jun;28(6):1717-1722. doi: 10.1681/ASN.2016060651. Epub 2017 Jan 3. PMID 28049648
- [Background] Nigwekar SU, Zhao S, Wenger J, Hymes JL, Maddux FW, Thadhani RI, Chan KE. A Nationally Representative Study of Calcific Uremic Arteriolopathy Risk Factors. J Am Soc Nephrol. 2016 Nov;27(11):3421-3429. doi: 10.1681/ASN.2015091065. Epub 2016 Apr 14. PMID 27080977
- [Background] Cozzolino M, Mangano M, Galassi A, Ciceri P, Messa P, Nigwekar S. Vitamin K in Chronic Kidney Disease. Nutrients. 2019 Jan 14;11(1):168. doi: 10.3390/nu11010168. PMID 30646590
- [Derived] D Shirsat P, Sonavane K, Botana LR, Sachdeva B. Calciphylaxis in the Upper GI Tract in an ESRD Patient: An Atypical Presentation and Review of Literature. Case Rep Nephrol. 2025 Dec 11;2025:3967671. doi: 10.1155/crin/3967671. eCollection 2025. PMID 41472909
- [Derived] Krishnasamy R, Jardine MJ; BEAT-Calci Trialists. Adaptive Designs for Clinical Trials in Nephrology. J Am Soc Nephrol. 2025 Jan 1;36(1):147-149. doi: 10.1681/ASN.0000000000000497. Epub 2024 Aug 26. No abstract available. PMID 39186385
- See also: Related Info — http://kidneyresearchcenter.mgh.harvard.edu/research